CLINICAL TRIAL: NCT05592106
Title: Comparing the Value of the Circular Region-of-interest- and Whole-liver Histogram-based Analysis on Gd-EOB-DTPA-enhanced T1 Map for Predicting Postoperative Liver Failure
Brief Title: Gd-EOB-DTPA-enhanced T1 Map for Predicting Postoperative Liver Failure
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2021-271
Record Dates: First submitted 2022-10-20; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Liver Failure
Keywords: Gd-EOB-DTPA; hepatectomy; liver failure; magnetic resonance imaging
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PHLF group and non-PHLF group: group with and without PHLF
  Interventions: Diagnostic Test: T1 mapping on gadoxetic acid-enhanced MRI

INTERVENTIONS:
Diagnostic Test: T1 mapping on gadoxetic acid-enhanced MRI — All subjects underwent 1.5T Gd-EOB-DTPA-enhanced MRI including pre-contrast and hepatobiliary-phase T1 mapping.

SUMMARY:
Researchers designed this study to compare the value of the conventional circular region-of-interest (ROI) and whole-liver histogram-based analysis on gadoxetic acid disodium (Gd-EOB-DTPA)-enhanced T1 map for predicting postoperative liver failure (PHLF). Researchers collected and analyzed the data of patients who underwent partial hepatectomy for focal liver lesions. Researchers drew circular ROIs on Gd-EOB-DTPA-enhanced T1 maps to get the mean T1 values. Researchers used a multiparametric analysis software to get histogram parameters. Then researchers compared the differences of these parameters between the PHLF group and non-PHLF group.

DETAILED DESCRIPTION:
The objective of this study is to compare the value of the circular region-of-interest (ROI) and whole-liver histogram-based analysis on gadoxetic acid disodium (Gd-EOB-DTPA)-enhanced T1 map for predicting postoperative liver failure. Forty patients who underwent partial hepatectomy for focal liver lesions were retrospectively analyzed. All subjects underwent 1.5T Gd-EOB-DTPA-enhanced MRI including pre-contrast and hepatobiliary-phase T1 mapping. Patients were divided into two groups with (16 patients) and without (24 patients) postoperative liver failure according to the criteria established by the International Study Group for Liver Surgery (ISGLS). T1 values before enhancement (T1pre) and in the hepatobiliary phase (T1HBP) were measured by outlining a circular ROI on the axial T1 maps. The reduction rate of T1 relaxation time (rrT1) = (T1 pre - T1HBP) / T1 pre. The whole-liver histogram analysis was performed using the prototype MR Multiparametric Analysis software (Siemens Healthcare, Erlangen, Germany). Differences of the circular ROI-based mean values and the histogram parameters between the two groups were compared. The receiver operating characteristic curve (ROC) was plotted. The circular ROI-based mean values and the histogram parameters for predicting PHLF was assessed by the area under the curve (AUC).

ELIGIBILITY:
Inclusion Criteria:

1. underwent liver resection; 2. underwent gadoxetic acid-enhanced MRI including, T1 mapping before and 20 minutes after gadoxetic acid administration within four weeks before the surgery ; 3. had an international normalized ratio (INR) and bilirubin examination on or after postoperative day five.

Exclusion Criteria:

1. patients who had undergone non-resection treatment, including chemotherapy, radiofrequency ablation, percutaneous ethanol injection, or transarterial chemoembolization; 2. patients whose images had severe respiratory motion artifacts.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the study group comprised 40 patients with an age range of 28 - 83 years (mean age, 58 years).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
postoperative liver failure | March, 2016- March, 2018
  increased INR and concomitant hyperbilirubinemia, according to the normal cut-off levels defined by the local laboratory on or after postoperative day five

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No